CLINICAL TRIAL: NCT00455312
Title: Hematopoietic Stem Cell Transplant For Patients With Dyskeratosis Congenita and Severe Aplastic Anemia
Brief Title: Stem Cell Transplant (SCT) for Dyskeratosis Congenita or SAA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT2006-06; 0612M98727 (Other: Institutional Review Board, University of Minnesota)
Record Dates: First submitted 2007-03-30; First posted 2007-04-03 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Dyskeratosis Congenita; Aplastic Anemia
Keywords: Dyskeratosis Congenita; Hematopoietic Stem Cell Transplantation; Severe Aplastic Anemia
MeSH Terms: conditions — Dyskeratosis Congenita; Anemia, Aplastic | interventions — Alemtuzumab; Cyclophosphamide; fludarabine; fludarabine phosphate; Whole-Body Irradiation; Radiotherapy; Stem Cell Transplantation; Bone Marrow Transplantation; Antilymphocyte Serum; thymoglobulin; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with DC (Experimental): Patients with dyskeratosis congenita (DC). Patients are treated with alemtuzumab (Campath 1H), Cyclophosphamide, Fludarabine, total body irradiation and stem cell transplantation.
  Interventions: Drug: Campath 1H; Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: Total Body Irradiation; Procedure: Stem Cell Transplantation
- Patients with SAA (Experimental): Patients with severe aplastic anemia (SAA). Patients are treated with alemtuzumab (Campath 1H), Cyclophosphamide, Fludarabine, antithymocyte globulin, total body irradiation and stem cell transplantation.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: Total Body Irradiation; Procedure: Stem Cell Transplantation; Drug: antithymocyte globulin; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Campath 1H — 10, 9, 8, 7, and 6 days before transplant subjects will be given 1 dose of campath 1H given via catheter (0.2 mg/kg over 2 hours).
  Other Names: Alemtuzumab
  Arms: Patients with DC
Drug: Cyclophosphamide — 7 days before the transplant, 1 dose of cyclophosphamide is given via catheter (50mg/kg IV over 2 hours).
  Other Names: Cytoxan
Drug: Fludarabine — 6, 5, 4, 3, and 2 days before the transplant, 1 dose fludarabine is given via catheter (40 mg/kg IV over 1 hour)
  Other Names: Fludara
Procedure: Total Body Irradiation — 1 day before the transplant one dose (200 cGy) of total body irradiation is given
  Other Names: Radiation therapy, therapeutic radiation
Procedure: Stem Cell Transplantation — Infusion of stem cells on Day 0.
  Other Names: Bone Marrow Transplant
Drug: antithymocyte globulin — ATG (rabbit) 3 mg/kg for 3 days.
  Other Names: Atgam; Thymoglobulin; ATG
  Arms: Patients with SAA
Drug: Methylprednisolone — 2mg/kg IV is given before each dose of antithymocyte globulin (ATG).
  Arms: Patients with SAA

SUMMARY:
Transplantation with stem cells is a standard therapy in many centers around the world. Previous experience with stem cell transplantation therapy for leukemias, lymphomas, other cancers, aplastic anemia and other non-malignant diseases, has led to prolonged disease-free survival or cure for some patients. However, the high doses of pre-transplant radiation and chemotherapy drugs used, and the type of drugs used, often cause many side effects that are intolerable for some patients. Slow recovery of blood counts is a frequent complication of high dose pre-transplant regimens, resulting in a longer period of risk for bleeding and infection plus a longer time in the hospital.

Recent studies have shown that using lower doses of radiation and chemotherapy (ones that do not completely kill all of the patient's bone marrow cells) before blood or bone marrow transplant, may be a better treatment for high risk patients, such as those with Dyskeratosis Congenita (DC) or Severe Aplastic Anemia(SAA). These low dose transplants may result in shorter periods of low blood counts, and blood counts that do not go as low as with traditional pre-transplant radiation and chemotherapy. Furthermore, in patients with Dyskeratosis Congenita or SAA, the stem cell transplant will replace the blood forming cells with healthy cells.

It has recently been shown that healthy marrow can take and grow after transplantation which uses doses of chemotherapy and radiation that are much lower than that given to patients with leukemia. While high doses of chemotherapy and radiation may be necessary to get rid of leukemia, this may not be important to patients with Dyskeratosis Congenita or SAA. The purpose of this research is to see if this lower dose chemotherapy and radiation regimen followed by transplant is a safe and effective treatment for patients with Dyskeratosis Congenita or SAA.

DETAILED DESCRIPTION:
This is an open label, single arm, phase II clinical trial designed to evaluate the safety and efficacy of the treatment regimen. Efficacy will be measured by long-term engraftment of the transplanted cells.The primary endpoint of neutrophil engraftment is defined as an absolute neutrophil count (ANC) >5 x 108/L (first of three consecutive laboratory measurements on different days) with at least 10% donor cells by day 100. We will evaluate the proportion of success (P) and its 95% confidence interval (CI) for the entire group. The null hypothesis of 90% engraftment will be rejected if 4 or more patients fail to engraft out of 15 evaluable patients. The secondary endpoints of regimen related mortality, acute and chronic graft-versus-host disease (GVHD) and secondary malignancies will be estimated by cumulative incidence treating non-event deaths as a competing risk. Survival will be estimated by Kaplan-Meier methods. Immune reconstitution will be summarized with descriptive statistics.

SAA and DC arms will be analyzed separately.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dyskeratosis congenita (DC) or severe aplastic anemia (SAA) 0-70 years of age with an acceptable hematopoietic stem cell (HSC) donor

  * HSC source

    * Human leukocyte antigen (HLA) identical or 1 antigen mismatched sibling or other relative eligible to donate bone marrow (BM), umbilical cord blood (UCB) or mobilized peripheral blood (PB) at cell doses that meet current institutional standards.
    * HLA identical or up to a 1 antigen mismatched unrelated donor.
    * Two units of unrelated umbilical cord blood (UCB) that are (a) up to 2 HLA antigens mismatched to the patient (b) up to 2 HLA antigens mismatched to each other, (c) minimum cell dose of ≥ 3.5 x 10^7 nucleated cells/kg and optimal cell dose ≥ 5 x 10^7 nucleated cells/kg.
    * If two units are not available: single unrelated UCB unit selected according to Minnesota Bone Marrow Transplant (BMT) program guidelines
  * Disease Characteristics for DC (both of the following):

    * Evidence of BM failure:

      * Requirement for red blood cell and/or platelet transfusions,
      * Requirement for granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) or erythropoietin, or
      * Refractory cytopenias defined as two out of three: platelets <40,000/microliter (uL) or transfusion dependent, Absolute neutrophil count <500/uL without hematopoietic growth factor support, Hemoglobin <9g/uL or transfusion dependent
    * Diagnosis of DC:

      * A triad of mucocutaneous features: oral leukoplakia, nail dystrophy, abnormal reticular skin hyperpigmentation.
      * Or one of the following: Short telomeres (under a research study), Dyskerin mutation, Telomerase RNA (TERC) mutation
  * Disease Characteristics for SAA (both of the following):

    * Evidence of BM failure:

      * Refractory cytopenia defined by bone marrow cellularity <25-50% (with < 30% residual hematopoietic cells)
    * Diagnosis of SAA:

      * Refractory cytopenias defined as two out of three: Platelets <20,000/uL or transfusion dependent, Absolute neutrophil count <500/uL without hematopoietic growth factor support, Absolute reticulocyte count <20,000/uL
  * Patients with early myelodysplastic features.
  * Patients with or without clonal cytogenetic abnormalities.

Patient Exclusion Criteria:

* Patients with one or more of the following:

  * Decompensated congestive heart failure; left ventricular ejection fraction <35%
  * Acute hepatitis or evidence of moderate or severe portal fibrosis or cirrhosis on biopsy
  * Carbon Monoxide Diffusing Capacity (DLCO) <30% predicted, and oxygen requirement
  * Glomerular filtration rate (GFR) <30% predicted
  * Pregnant or lactating female
  * Active serious infection whereby patient has been on intravenous antibiotics for at least one week prior to study entry. Any patient with AIDS or HIV seropositivity. If recent mold infection e.g. Aspergillus - must have >30 days of appropriate treatment before HSC transplantation and infection must be controlled and cleared by the Infectious Disease consultant.
  * Cannot receive total body irradiation (TBI) due to prior radiation therapy
  * Diagnosis of Fanconi anemia based on diepoxybutane (DEB).
  * DC patients with advanced myelodysplastic syndrome (MDS) or acute myeloid leukemia with >30 blasts.
  * History of non hematopoietic malignancy within 2 years except resected basal cell carcinoma or treated carcinoma in situ.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-08; Primary Completion 2015-03 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Tolar, M.D., Ph.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Dietz AC, Orchard PJ, Baker KS, Giller RH, Savage SA, Alter BP, Tolar J. Disease-specific hematopoietic cell transplantation: nonmyeloablative conditioning regimen for dyskeratosis congenita. Bone Marrow Transplant. 2011 Jan;46(1):98-104. doi: 10.1038/bmt.2010.65. Epub 2010 Apr 12. PMID 20383216

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With SAA: Patients with severe aplastic anemia (SAA). Patients are treated with alemtuzumab (Campath 1H), Cyclophosphamide, Fludarabine, antithymocyte globulin (ATG), total body irradiation and stem cell transplantation.
  Cyclophosphamide: 7 days before the transplant, 1 dose of cyclophosphamide is given via catheter (50mg/kg IV over 2 hours).
  Fludarabine: 6, 5, 4, 3, and 2 days before the transplant, 1 dose fludarabine is given via catheter (40 mg/kg IV over 1 hour)
  Total Body Irradiation: 1 day before the transplant one dose (200 cGy) of total body irradiation is given
  Stem Cell Transplantation: Infusion of stem cells on Day 0.
  antithymocyte globulin: ATG (rabbit) 3 mg/kg for 3 days.
  Methylprednisolone: 2mg/kg IV is given before each dose of ATG.
Period: Overall Study
Arm/Group | Patients With DC | Patients With SAA
Started | 15 | 21
Completed | 15 | 20
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Patients With SAA: Patients with severe aplastic anemia (SAA). Patients are treated with alemtuzumab (Campath 1H), Cyclophosphamide, Fludarabine, antithymocyte globulin, total body irradiation and stem cell transplantation.
  Cyclophosphamide: 7 days before the transplant, 1 dose of cyclophosphamide is given via catheter (50mg/kg IV over 2 hours).
  Fludarabine: 6, 5, 4, 3, and 2 days before the transplant, 1 dose fludarabine is given via catheter (40 mg/kg IV over 1 hour)
  Total Body Irradiation: 1 day before the transplant one dose (200 cGy) of total body irradiation is given
  Stem Cell Transplantation: Infusion of stem cells on Day 0.
  antithymocyte globulin: ATG (rabbit) 3 mg/kg for 3 days.
  Methylprednisolone: 2mg/kg IV is given before each dose of ATG.
- Total: Total of all reporting groups
Arm/Group | Patients With DC | Patients With SAA | Total
Number analyzed (Participants) | 15 | 21 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 15 | 21
  Between 18 and 65 years | 9 | 5 | 14
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 16
  Male | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Neutrophil Engraftment
Description: Defined as an absolute neutrophil count (ANC) >5 x 10^8/L (first of three consecutive laboratory measurements on different days) with at least 10% donor cells by day 100. Demonstrate sustained engraftment after a fludarabine based preparative regimen in patients with dyskeratosis congenita followed by hematopoietic cell transplantation.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With DC | Patients With SAA
Number analyzed (Participants) | 15 | 20
Participants | 15 | 20

2. Secondary Outcome: Incidence of Regimen Related Mortality at 100 Days
Description: all deaths without previous relapse or progression
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With DC | Patients With SAA
Number analyzed (Participants) | 15 | 21
Participants | 1 | 2

3. Secondary Outcome: Incidence of Chronic GVHD
Description: Chronic Graft-Versus-Host Disease is a severe long-term complication created by infusion of donor cells into a foreign host.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With DC | Patients With SAA
Number analyzed (Participants) | 15 | 21
Participants | 0 | 0

4. Secondary Outcome: Incidence of Chronic GVHD
Description: as for outcome 3
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With DC | Patients With SAA
Number analyzed (Participants) | 15 | 21
Participants | 1 | 2

5. Secondary Outcome: Incidence of Late Secondary Malignancies
Description: Defined as patients who have a secondary malignancy (cancer) occurring.
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With DC | Patients With SAA
Number analyzed (Participants) | 15 | 21
Participants | 0 | 4

6. Secondary Outcome: Incidence of Grade 2-4 Acute Graft Versus Host Disease (GVHD)
Description: Acute Graft-Versus-Host Disease is a severe short-term complication created by infusion of donor cells into a foreign host.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With DC | Patients With SAA
Number analyzed (Participants) | 15 | 21
Participants | 1 | 0

7. Secondary Outcome: Incidence of Grade 3-4 Acute Graft Versus Host Disease (GVHD)
Description: as for outcome 6
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With DC | Patients With SAA
Number analyzed (Participants) | 15 | 21
Participants | 0 | 0

8. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time from date of transplant to date of death or censored at the date of last documented contact for patients still alive.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With DC | Patients With SAA
Number analyzed (Participants) | 15 | 21
Participants | 14 | 19

9. Secondary Outcome: Overall Survival
Description: as for outcome 8
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With DC | Patients With SAA
Number analyzed (Participants) | 15 | 21
Participants | 12 | 19

10. Secondary Outcome: Incidence of Pulmonary Complications
Description: Defined as patients who exhibit a pulmonary (lung) adverse event.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With DC | Patients With SAA
Number analyzed (Participants) | 15 | 21
Participants | 3 | 3

ADVERSE EVENTS:
Arm/Group | Patients With DC | Patients With SAA
Serious Adverse Events (participants affected / at risk) | 2/15 | 1/21
Other Adverse Events (participants affected / at risk) | 15/15 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With DC (N=15) | Patients With SAA (N=21)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Intracranial Hemorrhage (Nervous system disorders) | 1 | 0
Pulmonary Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With DC (N=15) | Patients With SAA (N=21)
Acute Brain Infarction (Nervous system disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1
Acute Pancreatitis (Gastrointestinal disorders) | 0 | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Aseptic/Avascular Necrosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Blood Infection (Infections and infestations) | 10 | 14
Bone Marrow Biopsy Site Infection (Infections and infestations) | 1 | 0
Bone Marrow Infection (Infections and infestations) | 0 | 1
Capillary Leak Syndrome (Vascular disorders) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 2
Coagulopathy (Investigations) | 0 | 1
Colitis (Infections and infestations) | 0 | 1
Congestive Heart Failure (Cardiac disorders) | 1 | 0
Cystitis (Renal and urinary disorders) | 2 | 3
Cytopenias (Blood and lymphatic system disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 1
Ear Infection (Infections and infestations) | 1 | 0
Early Small Bowel Obstruction vs. Ileus (General disorders) | 1 | 0
Epstein Barr Virus Infection (Infections and infestations) | 0 | 1
Erythema at Central Line Site (Skin and subcutaneous tissue disorders) | 0 | 1
Erythroid Aplasia (Blood and lymphatic system disorders) | 0 | 1
Eye Infection (Infections and infestations) | 1 | 0
Fever (General disorders) | 0 | 1
Fever with Chills (General disorders) | 0 | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Gallstones (Hepatobiliary disorders) | 0 | 1
GI Bleed (Gastrointestinal disorders) | 3 | 2
GI Infection (Infections and infestations) | 1 | 4
Hemorrhagic Pancreatitis (Gastrointestinal disorders) | 0 | 1
Herpes Zoster (Infections and infestations) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 4 | 8
Hypogonadism (Endocrine disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infection at Central Line Site (Infections and infestations) | 0 | 1
Labia Infection (Infections and infestations) | 1 | 0
Low Reticulocyte Count (Blood and lymphatic system disorders) | 0 | 1
Lung Collapse (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Meningitis (Nervous system disorders) | 1 | 0
Multi Organ Failure (General disorders) | 1 | 0
Nasal Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Anorexia (Gastrointestinal disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 1 | 1
Brain Lesion, Nonspecific (Nervous system disorders) | 0 | 1
Nose Bleeds (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Otomastoiditis (Ear and labyrinth disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 1 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 | 10
Intra-Abdominal Infection, Unconfirmed (Infections and infestations) | 0 | 1
Pulmonary Hypertension (Cardiac disorders) | 0 | 1
Post Transplant Lymphoproliferative Disease (Blood and lymphatic system disorders) | 0 | 1
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pustular Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Pyelocaliectasis (Renal and urinary disorders) | 0 | 1
Renal Injury Requiring Dialysis (Renal and urinary disorders) | 0 | 1
Respiratory Infection (Infections and infestations) | 1 | 3
Retinal Hemorrhage (Eye disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Skin Infection (Infections and infestations) | 2 | 3
Spongiotic Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Tonsilar Infection (Infections and infestations) | 0 | 1
Transaminitis (Investigations) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 2 | 0
Vaginal Infection (Infections and infestations) | 0 | 1
Veno-Occlusive Disease (Hepatobiliary disorders) | 0 | 1
Vocal Fold Erythema and Leukoplakia (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No